CLINICAL TRIAL: NCT04613063
Title: Proximal Intestinal Obstruction Syndrome (PIOS) in a Patient With Cystic Fibrosis: A New Syndrome
Status: Completed | Type: Observational
Sponsor: Tecnologico de Monterrey (Other)
Responsible Party: Sponsor
Other Study IDs: I1568Z
Record Dates: First submitted 2020-10-21; First posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Cystic Fibrosis; Bowel Obstruction; Distal Intestinal Obstruction Syndrome
MeSH Terms: conditions — Cystic Fibrosis; Intestinal Obstruction | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Diagnostic laparoscopy — A diagnostic laparoscopy was performed where a dilated jejunum was encountered with impaction of fecal content. Surgery was converted to open surgery, where a longitudinal enterotomy of 5 cm after the transition zone was created, evacuating manually the fecal material with mucous secretion.

SUMMARY:
A case of a patient with cystic fibrosis with bowel obstruction due to a proximal intestinal obstruction syndrome (PIOS) is presented.This syndrome can be diagnosed with the DIOS definition, with the only distinction of a more proximal location in the gastrointestinal tract, such as the stomach, the duodenum, or the jejunum.

DETAILED DESCRIPTION:
Distal Intestinal Obstruction Syndrome is a rare complication in cystic fibrosis patients characterized by the accumulation of viscid fecal material, combined with sticky mucous secretions located in the distal ileum, adhered to the intestinal wall. Only few cases have been reported in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Adult >18 years
* Cystic fibrosis
* Bowel obstruction

Exclusion Criteria:

* Pediatric patient <18 years
* Unknown cause of bowel obstruction

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 45 years old patient with cystic fibrosis
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
Bowel obstruction in a patient with cystic fibrosis | 3-6 days
  A 45 year old patient with cystic fibrosis presented with bowel obstruction. Image studies were performed, without identifying a specific cause of the bowel obstruction. The patient was transferred to surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Escuela Nacional de Medicina, Tecnologico de Monterrey, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No